CLINICAL TRIAL: NCT04596527
Title: Diagnostic Performance of 18F-FMPP PET Myocardial Perfusion Imaging in the Detection of Coronary Artery Disease: A Comparative Study With 13N-Ammonia PET
Brief Title: 18F-FMPP PET MPI in the Detection of Coronary Artery Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZS-2514
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FMPP PET MPI (following off-study 13N-ammonia PET MPI) (Experimental): Imaging Procedure: 18F-FMPP PET Day 1: All subjects will receive rest and stress IV boluses of 18F-FMPP injections in a large peripheral vein. The dosages of 18F-FMPP Injection administered at rest and during stress conditions are 2.5 mCi and 6.0 mCi for an individual subject. Rest or stress PET imaging will be acquired for 20 minutes. The pharmacological stress will utilize ATP as the stressor.
  Imaging Procedure: 13N-Ammonia PET All subjects will receive 2 IV boluses of 13N-ammonia Injection in a large peripheral vein: 1 at rest and 1 during stress. The dosages of 13N-ammonia Injection administered at rest and during stress conditions is 20mCi and 20 mCi for an individual subject. Rest or stress PET imaging will be acquired for 20 minutes. The pharmacological stress will utilize ATP as the stressor.
  Interventions: Drug: 18F-FMPP

INTERVENTIONS:
Drug: 18F-FMPP — 18F-FMPP were injected into the patients at rest (2.5 mCi) and during stress (6.0 mCi) for an individual subject before PET/CT scans.
  Other Names: XTR004

SUMMARY:
18F-FMPP is a novel PET myocardial perfusion imaging (MPI) tracer which targets to mitochondria complex I (MC-I). Preclinical animal studies have shown that its uptake is highly uniform and long in the heart and rather low in the liver. It may be a promising tracer for myocardial perfusion imaging. In addition, as a myocardial PET tracer, it is capable of quantifying absolute myocardial blood flow. Thus this prospective and open-label study is going to evaluate the diagnosis performance of 18F-FMPP PET MPI in suspected or known CAD patients who will be referred for invasive coronary angiography (ICA).

DETAILED DESCRIPTION:
PET myocardial perfusion imaging (MPI) can provide not only qualitative images, but also absolute quantitation of myocardial blood flow (MBF) in the unit of ml/min/g to facilitate the early diagnosis of coronary disease (CAD). It can be more beneficial for patients with three-vessel disease, microvascular disease or obesity. At present, the diagnostic capability of 13N-ammonia PET MPI has been well studied, but its clinical usability is largely limited by short half-life. 18F-labeled MPI tracer (18F-FMPP) is a new type of PET tracer for MPI. Preclinical studies showed that 18F-FMPP has important characteristics such as high myocardial retention and low background uptake of adjacent organs, which may be a more ideal drug for PET MPI toward routine clinical utilization. Our study will assess the safety profile, image quality and diagnostic performance of 18F-FMPP PET in detection of CAD by using invasive coronary angiography as the reference standard. In addition, the investigators will further compare the diagnostic performance of 18F-FMPP PET MPI with that of 13N-ammonia PET MPI.

ELIGIBILITY:
Inclusion Criteria:

* The subject has read, signed, and dated an informed consent form (ICF) prior to any study procedures being performed.
* At the time of enrolment, the subject has been scheduled via written documentation to undergo an ICA for the assessment of CAD.
* The subject at least has one or multiple risk factors for coronary heart disease, including hypertension, hyperlipidemia, hyperglycemia, smoking, family history, obesity, post-menopause.
* The subject presents typical symptoms for CAD such as dyspnea, chest tightness and chest pain.
* The subject is male or is a nonpregnant, nonlactating female who is either surgically sterile or is post-menopausal.
* The subject is able and willing to comply with all study procedures as described in the protocol.

Exclusion Criteria:

* Patients who are pregnant, may possibly be pregnant, or wish (including their partners) to become pregnant during the study period, or are lactating.
* Patients incapable of undergoing pharmacological cardiac stress testing.
* Patients who have a current illness or pathology that, in the opinion of the investigator, would pose a significant safety risk for the patient during cardiac stress testing.
* Documented history of heart failure and/or cardiomyopathy and/or prior LV ejection fraction (LVEF <50%).
* Patients whose images quality can not meet the requirements.
* Patients who are not suitable to participate in the trial according to researchers.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
The evaluation of diagnostic performance of 18F-FMPP PET MPI in the detection of CAD | through study completion, an average of 2 years
  Defined by invasive coronary angiography in patients with suspected or known CAD

SECONDARY OUTCOMES:
Diagnostic rate of 18F-FMPP MPI in CAD patients | through study completion, an average of 2 years
  Diagnostic efficacy of 18F-FMPP PET MPI compared with 13N-ammonia PET MPI in the detection of CAD in patients with suspected or known CAD.
  Qualitative PET MPI alone. Absolute MBF quantitation alone. Added value of MBF quantitation
Number of Participants with Adverse events | through study completion, an average of 2 years
  Number of participants and type of adverse events as a measure of safety
good quality rate of images | through study completion, an average of 2 years
  18F-FMPP and 13N-ammonia PET MPI images

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking union medical college hospital, Beijing, Dongcheng, China

IPD SHARING:
Plan to Share IPD: No